CLINICAL TRIAL: NCT05842668
Title: Investigation of the Effect of Virtual Glasses Used During Extracorporeal Shock Wave Lithotripsy-ESWL on Patient's Pain and Comfort Level: A Randomized Controlled Study
Brief Title: Effect of Virtual Glasses on Pain and Comfort During ESWL
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The run could not be started
Sponsor: Akdeniz University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Seda Cansu Yeniğün, Lecturer, Akdeniz University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Lecturer-11412
Record Dates: First submitted 2023-04-20; First posted 2023-05-06 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Extracorporeal Shock Wave Lithotripsy; Lithotripsy
Keywords: ESWL; Pain; comfort level; virtual glasses
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ESWL Group (Experimental)
  Interventions: Behavioral: ESWL Group
- Control Group (No Intervention)

INTERVENTIONS:
Behavioral: ESWL Group — Increasing comfort and reducing pain during ESWL
  Arms: ESWL Group

SUMMARY:
The aim of this study is to examine the effect of virtual glasses application on the patient's pain and comfort level during ESWL.

The data obtained in the research will be analyzed using the SPSS 23.0 "Statistical Package for Social Sciences" for Windows program. Descriptive statistical methods when evaluating data; number, percentage, mean, frequency, standard deviation will be used. As hypothesis tests, analysis will be made with Mann Whitney U, student t test, and chi-square tests. The findings will be interpreted with a significance level of 0.05 at the 95% confidence interval.

DETAILED DESCRIPTION:
After obtaining the permission of the ethics committee and institution of the study, the researcher will go to the clinic and introduce himself to the patient who is admitted to undergo ESWL procedure and explain the purpose of the research. Informed consent will be obtained from patients who volunteered to participate in the study. The data on the socio-demographic characteristics of the patients in the patient introduction form will be interviewed face-to-face with the patient, and the data on the clinical characteristics of the patients will be recorded from the patient file. Data will be collected from the first patient who will undergo the ESWL procedure. Pain with VAS and comfort level with General comfort scale will be checked 5-10 minutes before the procedure. According to the randomization, the patient in the virtual glasses group will first be explained to the patient by the researcher that he will wear the glasses for 30 minutes during the procedure and watch the video. When the 30 minutes are up, the patient will be informed by the researcher and the glasses will be removed. No intervention will be performed on the patient in the control group. The first patient will go to the operation room. Patients in the virtual glasses group will use the virtual glasses for 30 minutes after the patient goes to the operating table and the preparation is completed. No intervention will be performed on the patient in the control group. All patient groups will be checked for pain with VAS and comfort level with general comfort scale 30 minutes after the end of the procedure. At the end of the procedure, the patient will come to the service. No intervention will be done to the patients in the control group, and the routine care protocol of the clinic will be applied.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older,
* Absence of hearing and perception problems,
* Absence of any visual impairment,
* ESWL procedure will be performed for the first time,

Exclusion Criteria:

* Using any analgesic or anxiolytic before the procedure,
* Having a psychiatric disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-03-16 (Estimated)

PRIMARY OUTCOMES:
Comfort Score | 5-10 minutes before ESWL
  The response patterns of the scale, which consists of positive and negative items, are given in a mixed form. A high score for positive items (4) indicates high comfort, a low score (1) indicates low comfort, and a low score (1 point) for negative items indicates high comfort, and a high score (4 points) indicates low comfort. While evaluating the scale, the negative scores obtained are reverse coded and added together with the positive items. The maximum total score that can be obtained from the scale is 192, and the minimum total score is 48.
Pain Score (Visual analog Score) | 5-10 minutes before ESWL
  Grading is made with a 10 cm long horizontal or vertical ruler on the scale and "0" means no pain and "10" means the most severe pain.
  The patient marks the intensity of pain he feels on the ruler. If the marked value is between 1-4, it indicates mild pain, between 5-6 indicates moderate pain, and between 7-10 indicates severe pain.
  In the application, the patient was asked to mark the intensity of pain he felt on the ruler and the value was measured and recorded.

SECONDARY OUTCOMES:
Comfort Score | 15 minutes after ESWL
  The response patterns of the scale, which consists of positive and negative items, are given in a mixed form. A high score for positive items (4) indicates high comfort, a low score (1) indicates low comfort, and a low score (1 point) for negative items indicates high comfort, and a high score (4 points) indicates low comfort. While evaluating the scale, the negative scores obtained are reverse coded and added together with the positive items. The maximum total score that can be obtained from the scale is 192, and the minimum total score is 48.
Pain Score (Visual analog Score) | 15 minutes after ESWL
  Grading is made with a 10 cm long horizontal or vertical ruler on the scale and "0" means no pain and "10" means the most severe pain.
  The patient marks the intensity of pain he feels on the ruler. If the marked value is between 1-4, it indicates mild pain, between 5-6 indicates moderate pain, and between 7-10 indicates severe pain.
  In the application, the patient was asked to mark the intensity of pain he felt on the ruler and the value was measured and recorded.

IPD SHARING:
Plan to Share IPD: No